CLINICAL TRIAL: NCT01517438
Title: Effects of Serotonin Inhibitors on Patient-controlled Analgesia Related Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Department of Anesthesiology and Pain Medicine, Seoul National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: ramosetron
Record Dates: First submitted 2012-01-17; First posted 2012-01-25 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Agitation
Keywords: agitation, desflurane, children
MeSH Terms: conditions — Psychomotor Agitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

INTERVENTIONS:
Behavioral: agitation — agitation score after desflurane anesthesia

SUMMARY:
ED50 of dexmedetomidine for prevention of emergence agitation after tonsillectomy or adenoidectomy in children

ELIGIBILITY:
Inclusion Criteria:

* tonsillectomy or adenoidectomy

Exclusion Criteria:

* development delay,
* CNS abnormality

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
agitation score | 30 minutes after postoperatuib
  agitation score